CLINICAL TRIAL: NCT00930878
Title: A Comparative Registry of the PROmus™, ENdeavor™ and CYpher™ Drug Eluting Coronary Stent Systems for the Treatment of Coronary Lesions
Brief Title: Comparative Registry of the PROmus™, ENdeavor™ and CYpher™ Drug Eluting Stents
Acronym: ProEnCy
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: S2213
Record Dates: First submitted 2008-03-26; First posted 2009-07-02 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Percutaneous Coronary Intervention
Keywords: registry; drug eluting coronary stent system; observational; prospective; open-label

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Promus: Patients intended to be treated with a Promus™ stent system
  Interventions: Device: Cardiac Stenting
- Endeavor: Patients intended to be treated with an Endeavor™ stent system (excluded the Endeavor™ Resolute™ stent)
  Interventions: Device: Cardiac Stenting
- Cypher: Patients intended to be treated with a Cypher™ stent system
  Interventions: Device: Cardiac Stenting

INTERVENTIONS:
Device: Cardiac Stenting — Drug Eluting stent

SUMMARY:
The purpose of this study is to collect real-life data of the Promus™ stent, the Cypher™ stent and the Endeavor™ stent in routine clinical practice, and compare outcomes.

DETAILED DESCRIPTION:
Boston Scientific is developing the present PROENCY registry to collect real world data with the Promus™ Stent and to compare outcomes to the Cypher™ and Endeavor™ stents.

All three stents have received CE Mark and are commonly used in Europe. All the data collected in this registry will be from patients treated according to the physician's choices, per Product Directions/Instructions for Use, per approved indications and per local standard of care.

The results from this registry will provide an understanding of the use and outcomes associated with the Promus™, the Endeavor™ and the Cypher™ stent systems in a real world setting.

ELIGIBILITY:
All the data collected in this registry will be from patients treated according to the physician's choices, per Product Directions/Instructions for Use, per approved indications and per local standard of care.

Inclusion Criteria:

* Per PROMUS or CYPHER or Endeavor DFU/IFU

PROMUS Indications:

* PROMUS™ Everolimus Eluting Coronary Stent System is indicated for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de novo native coronary artery lesions (length 28 mm) with a reference vessel diameter of 2.5 mm - 4.0 mm.

CYPHER Indications:

* CYPHER SELECT Sirolimus-eluting Coronary Stent is indicated for improving coronary luminal diameter in patients with symptomatic ischemic disease due to discrete de novo and in-stent restenotic lesions (length 30 mm) in native coronary arteries with a reference vessel diameter of 2.25 mm to 5.00 mm.

Endeavor Indications:

* Endeavor Stent is indicated for improving coronary luminal diameter and reducing restenosis in patients with symptomatic ischemic heart disease in de novo coronary artery lesions in native coronary arteries with a reference vessel diameter of 2.25 mm to 4.0 mm and a lesion length of < 27 mm.

Exclusion Criteria:

PROMUS Contraindications:

* Patients in whom anti-platelet and / or anti-coagulant therapy is contraindicated.
* Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Patients with a known hypersensitivity or contraindication to everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro - polymers may have an allergic reaction to this implant; therefore, the implant is not recommended for such patients.

CYPHER Contraindications:

* Patients in whom antiplatelet and/or anticoagulation therapy is contraindicated.
* Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon.
* Transplant patients.

Endeavor Contraindications:

* Patients with hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, drugs such as ABT-578, rapamycin, tacrolimus, sirolimus or similar drugs or any other analogue or derivative, cobalt, chromium, nickel, molybdenum, or contrast media.
* Patients in whom antiplatelet and/or anticoagulation therapy is contraindicated.
* Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients eligible and planned for percutaneous coronary intervention (PCI) with any of the three stents and willing to give consent to allow for collection of their clinical data. Patients also need to express willingness to comply with all standard of care follow-up evaluations and medical therapies.
Sampling Method: Probability Sample
Enrollment: 1934 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Rate of composite patient-oriented hierarchical Major Cardiac Events and its individual components (cardiac death, any Myocardial Infarction (MI) and Target Vessel Revascularisation (TVR) as classified by an External Medical Monitoring Committee. | at 12-month post index procedure

SECONDARY OUTCOMES:
Technical Success, Stent deliverability, Rate of composite stent-oriented hierarchical Major Cardiac Events and its individual components, TVR rates, TLR rates, Rate of all death, Rate of stent thrombosis | at 6 and/or 12 months post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Christian Hamm, MD, Principal Investigator — Kerckhoff-Klinik GmbH
Locations (1):
- Kerckhoff-Klinik GmbH, Bad Nauheim, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No